CLINICAL TRIAL: NCT02210650
Title: Randomized Controlled Trial Comparing Relapse Rates Between Standard Ureteroscopic Removal Of Ureteral Stone And Standard Removal With Additional Ureterorenic Clearing Of Non-Symptomatic Stones In The Kidney
Brief Title: Trial Comparing Relapse Rates Between Standard Ureteroscopic Removal Of Ureteral Stone And Standard Removal With Additional Ureterorenic Clearing Of Non-Symptomatic Stones In The Kidney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: University of Washington (Other); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01 DK 043881 Project 3; P01DK043881 (NIH)
Record Dates: First submitted 2014-08-01; First posted 2014-08-07 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Ureteral Stones, Kidney Stones
Keywords: kidney stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symptomatic stone removal (Other): Group 1 will receive the standard treatment of having only the symptomatic stone removed
  Interventions: Procedure: Symptomatic stone removal
- Asymptomatic kidney stones and symptomatic stone removed (Other): Group 2 will include the step of having the asymptomatic kidney stones removed in addition to the symptomatic stone
  Interventions: Procedure: Asymptomatic kidney stones and ureteral stone removed

INTERVENTIONS:
Procedure: Symptomatic stone removal — Symptomatic stone removal by the surgical procedures called Ureteroscopy or Percutaneous Nephrolithotomy
  Arms: Symptomatic stone removal
Procedure: Asymptomatic kidney stones and ureteral stone removed — Asymptomatic kidney stones and symptomatic stone removal by the surgical procedure called Ureteroscopy
  Arms: Asymptomatic kidney stones and symptomatic stone removed

SUMMARY:
Patients with a ureteral or kidney stone that causes symptoms, like pain, frequently have small kidney stones that don't cause symptoms. If these small kidney stones are determined to be asymptomatic (not causing any problems or pain), then most urologists will simply remove the symptomatic ureteral stone and leave the additional stones in the kidneys. However, symptomatic kidney stones started as small stones that didn't cause symptoms. This means that the small stones remaining in the patient's kidney may cause problems later. The purpose of our research is to test if removing small stones from the kidney prevents future stone episodes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo surgery (URS or PCNL) for a primary stone.
* Computed tomography (CT) exam within the 90-day pre-operative period
* Small (≤ 6mm) asymptomatic stones in visible on KUB or CT (i.e., calcium stones) in the contralateral kidney for a primary renal stone or ipsilateral kidney for primary ureteral stone.
* Recurrent (having had previous stones) or multiple (simultaneous bilateral stones) stones
* Able to give informed consent
* Age 21 years or older

Exclusion Criteria:

* Inability to give informed consent
* Age less than 21 years
* Stones not visible on KUB or CT
* Patients with systemic disease or renal anatomical disorders (RTA, primary hyperparathyroidism, sarcoidosis, enteric hyperoxaluria, medullary sponge kidney)
* Any condition (eg, psychiatric illness) or situation that, in the investigator's opinion, could put the
* subject at significant risk, confound the study results, or interfere significantly with the subject's
* participation in the study.
* Unwilling to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-11; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Relapse of stone disease on the study side | annually up to 5 years after stone removal surgery
  1. Radiological evidence of significant growth in the size of any pre-existing stone
  2. Return for stone removal surgery on the study side
  3. Passage of a stone with pain symptoms on the study side resulting in an emergency department visit

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — Indiana University Health
Locations (4):
- United States (4):
  - Indiana University Health, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - University of Washington Medical Center Department of Urology, Seattle, Washington
  - Veterans Administration Puget Sound Heath Care System, Seattle, Washington

REFERENCES:
- [Derived] Sorensen MD, Harper JD, Borofsky MS, Hameed TA, Smoot KJ, Burke BH, Levchak BJ, Williams JC Jr, Bailey MR, Liu Z, Lingeman JE. Removal of Small, Asymptomatic Kidney Stones and Incidence of Relapse. N Engl J Med. 2022 Aug 11;387(6):506-513. doi: 10.1056/NEJMoa2204253. PMID 35947709